CLINICAL TRIAL: NCT01355107
Title: Comparison of Selenium Levels in HCV- Infected Patients at Different Stages of Disease - a Pilot Trial
Brief Title: Comparison of Selenium Levels in HCV- Infected Patients at Different Stages of Disease
Status: Completed | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Collaborators: Biosyn (Industry)
Responsible Party: Principal Investigator, Dominik Bettinger, investigator, University Hospital Freiburg
Other Study IDs: HCC1; DRKS00000813 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2011-05-06; First posted 2011-05-17 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Hepatitis C; Liver Cirrhosis; Carcinoma, Hepatocellular
Keywords: selenium level measurement
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- chronic hcv, no liver cirrhosis, no HCC: patients with chronic hepatitis c- infection: no cirrhosis of the liver (= Desmet IV), no HCC - suspected lesion in the liver
- chronic hcv, liver cirrhosis, no HCC: patients with hcv- associated cirrhosis of the liver, but with no HCC - suspected lesions in the liver
- hcv-infection, HCC: patients with hcv- associated HCC

SUMMARY:
The incidence of hepatocellular carcinoma (HCC) is rising worldwide.One important etiology is a chronic inflammation due to hepatitis c (hcv) infection. Over the steps of a chronic inflammation over the stadium of cirrhosis of the liver it is possible that neoplastic nodules appear in the liver which can rise up to a HCC. In the pathogenesis of HCC oxidative stress seems to play an important role and as selenium is a key micronutrient in this process its levels could differ between the different stages of disease in hcv- infected patients. The aim of this trial is to examine these differences.

DETAILED DESCRIPTION:
The incidence of hepatocellular carcinoma (HCC) is rising worldwide. Almost all cases of HCC develop over clearly defined stages of chronic hepatic inflammation and cirrhosis of the liver which can be determined as an irreversible stage during this process. In the Western world excessive alcohol consumption and chronic infection with the hepatitis c virus (hcv) are frequent causes of chronic hepatocellular injury. As HCC is often diagnosed at advanced stages and therapeutic intervention possibilities are limited it becomes more and more necessary to search for prevention strategies to stop the development of HCC.

In the last years micronutrients such as selenium have reached the interests of oncologists. Several studies were able to show that there are often low selenium levels in patients with different tumors. Some epidemiologic studies showed that supplementation of selenium can decrease the incidence of some tumors.

Oxidative stress is meant to play an essential role in hepatocarcinogenesis and as selenium could decrease it, it may be possible that patients infected with the hepatitis c - virus show low selenium levels probably as a result of the chronic hepatic inflammation. Moreover there may be differences between the stages of disease namely chronic infection, cirrhosis of the liver and hepatocellular carcinoma. The aim of this trial is to determine these differences.

HCV- infected patients are enrolled in this trial. Three groups are formed: In Group 1 all HCV- infected patients with a chronic inflammation without cirrhosis of the liver and without HCC are summarized. in group 2 all HCV- infected patients with cirrhosis of the liver but without HCC are enrolled. In group 3 hcv- infected HCC- patients are summarized. In each group 10 patients should be enrolled, matched to age and other diseases. Blood samples are taken from these patients and selenium levels are measured.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic hepatitis c- infection: no cirrhosis of the liver (= Desmet IV), no HCC - suspected lesion in the liver
* patients with hcv- associated cirrhosis of the liver: - cirrhosis of the liver confirmed by ultrasound, CT/MRI imaging or biopsy, all child - stages
* patients with hcv- associated HCC: diagnosis of HCC according to the AASLD criteria, HCC has not been treated at the time of enrollment, all BCLC- /UICC- stages.
* for all three groups: diagnosis of the chronic hcv- infection with virus rna and serologic parameters (anti-hcv) and abnormal liver function for more than 6 months, no antiviral treatment during the last 6 months

Exclusion Criteria:

* application of dietary supplements
* excessive alcohol consumption
* all other etiologies leading to a liver injury
* patients with an acute-phase- reaction, SIRS or patients in intensive care units
* extrahepatic neoplasm
* rheumatic disease apart from hcv- associated immunologic phenomena
* diabetes mellitus I and II
* immunological diseases

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Whole blood samples are taken from inpatients and outpatients of our primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
measurement of selenium levels in hcv- infected patients | baseline
  measurement of selenium levels in whole blood samples

SECONDARY OUTCOMES:
selenium levels and inflammatory activity | baseline
  determination if there is a correlation between selenium levels and inflammatory activity
selenium levels and stage of HCC (BCLC, UICC) | baseline
  determination if there is a correlation between selenium levels and the stage of HCC (BCLC, UICC)
selenium levels and MELD(Na)score | baseline
  determination if there is a correlation between selenium levels and the MELD(Na)-score

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Spangenberg, Prof. Dr., Principal Investigator — University Medical Center Freiburg
Locations (1):
- University Medical Center Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Muecke R, Schomburg L, Buentzel J, Kisters K, Micke O; German Working Group Trace Elements and Electrolytes in Oncology. Selenium or no selenium--that is the question in tumor patients: a new controversy. Integr Cancer Ther. 2010 Jun;9(2):136-41. doi: 10.1177/1534735410367648. Epub 2010 May 11. PMID 20462857
- [Background] Brenneisen P, Steinbrenner H, Sies H. Selenium, oxidative stress, and health aspects. Mol Aspects Med. 2005 Aug-Oct;26(4-5):256-67. doi: 10.1016/j.mam.2005.07.004. PMID 16105679
- [Background] Shamberger RJ, Rukovena E, Longfield AK, Tytko SA, Deodhar S, Willis CE. Antioxidants and cancer. I. Selenium in the blood of normals and cancer patients. J Natl Cancer Inst. 1973 Apr;50(4):863-70. doi: 10.1093/jnci/50.4.863. No abstract available. PMID 4703775
- [Background] Sakoda LC, Graubard BI, Evans AA, London WT, Lin WY, Shen FM, McGlynn KA. Toenail selenium and risk of hepatocellular carcinoma mortality in Haimen City, China. Int J Cancer. 2005 Jul 1;115(4):618-24. doi: 10.1002/ijc.20937. PMID 15704105
- [Background] Yu MW, Horng IS, Hsu KH, Chiang YC, Liaw YF, Chen CJ. Plasma selenium levels and risk of hepatocellular carcinoma among men with chronic hepatitis virus infection. Am J Epidemiol. 1999 Aug 15;150(4):367-74. doi: 10.1093/oxfordjournals.aje.a010016. PMID 10453813
- [Background] Yu SY, Zhu YJ, Li WG, Huang QS, Huang CZ, Zhang QN, Hou C. A preliminary report on the intervention trials of primary liver cancer in high-risk populations with nutritional supplementation of selenium in China. Biol Trace Elem Res. 1991 Jun;29(3):289-94. doi: 10.1007/BF03032685. PMID 1726411
- [Background] Lin CC, Huang JF, Tsai LY, Huang YL. Selenium, iron, copper, and zinc levels and copper-to-zinc ratios in serum of patients at different stages of viral hepatic diseases. Biol Trace Elem Res. 2006 Jan;109(1):15-24. doi: 10.1385/BTER:109:1:015. PMID 16388099
- [Background] Navarro-Alarcon M, Lopez-Ga de la Serrana H, Perez-Valero V, Lopez-Martinez MC. Selenium concentrations in serum of individuals with liver diseases (cirrhosis or hepatitis): relationship with some nutritional and biochemical markers. Sci Total Environ. 2002 May 27;291(1-3):135-41. doi: 10.1016/s0048-9697(01)01088-9. PMID 12150433
- [Background] Martinez-Peinado M, Nogueras-Lopez F, Arcos-Cebrian A, Agil A, Navarro-Alarcon M. Serum selenium levels in cirrhotic patients are not influenced by the disease severity index. Nutr Res. 2010 Aug;30(8):574-8. doi: 10.1016/j.nutres.2010.08.004. PMID 20851312